CLINICAL TRIAL: NCT00746525
Title: Non-Invasive Brain Signal Training to Induce Motor Control Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Janis Daly, Director, Brain Rehabilitation Research Center, North Florida/South Georgia Veterans Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R01NS063275 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: stroke; motor learning; rehabilitation of upper extremity; functional electrical stimulation; FES; brain computer interface; BCI; coordination; motor control
MeSH Terms: conditions — Stroke | interventions — Brain-Computer Interfaces; 2-benzylidene-3-(cyclohexylamino)-2,3-dihydro-1H-inden-1-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Computer Interface Training Stroke Experimental Group (Experimental): Individuals in the stroke experimental group received treatment with BCI, FES, and motor learning targeted at their upper extremity motor deficits following stroke.
  Interventions: Other: Surface functional electrical stimulation (FES); Other: Motor learning; Other: Brain computer interface (BCI) training

INTERVENTIONS:
Other: Surface functional electrical stimulation (FES) — FES is a technique that electrically stimulates a muscle in a comfortable manner in order to contract the muscle. It uses an electrode placed on the surface of the skin. This study will use BCI, FES, and motor learning interventions to address upper extremity motor deficits following stroke.
Other: Motor learning — Motor learning is an exercise that uses movements needed for everyday tasks such as picking up a glass or opening a book. This study will use BCI, FES, and motor learning interventions to address upper extremity motor deficits following stroke.
Other: Brain computer interface (BCI) training — BCI training uses signals produced by the brain to help individuals with stroke move their weak arm. This study will use BCI, FES and motor learning interventions to address upper extremity motor deficits following stroke.

SUMMARY:
The purpose of this trial was to evaluate the benefits of combination motor learning training and brain computer interface training for restoring arm function in people with stroke. Our aim was to determine whether the surface-acquired brain signal (electroencephalography (EEG)) can feasibly be used as a neural feedback system to drive more normal motor function in stroke survivors.

DETAILED DESCRIPTION:
The financial burden and human suffering are devastating after stroke due to the lack of rehabilitation protocols that can restore normal brain and motor function. Conventional treatment does not restore normal motor function to many stroke survivors. The majority of available treatments are directed at the peripheral nervous system (arms/legs). Since stroke occurs in the brain and results in brain damage and dysfunction, a more direct approach may be to re-train the brain by directly treating the activation of brain signals that control movement.

The purposes of this study are to determine if motor learning, functional electrical stimulation (FES), and brain computer interface (BCI) training are beneficial for restoring arm function in people who have had a stroke, and to determine if the surface-acquired brain signal [electroencephalography (EEG)] can be re-trained to provide more normal motor function in stroke survivors. The primary purpose of this study is to determine the efficacy of the motor learning tasks in stroke recovery.

In the study, scientists will use two different and complimentary brain signal training components to restore more normal motor control of a motor task (elbow, wrist, or finger movement task). Specifically targeting, invoking, and training the surface-acquired EEG brain signal, and integrating brain signal training into motor learning training of upper limb motor tasks, may result in greater motor restoration when compared to a comprehensive motor learning intervention without EEG brain signal training.

Eight people who had a stroke were enrolled in the experimental group. They received brain signal training and comprehensive motor learning based therapy.

An additional 5 healthy adults were enrolled in order to study their ability to acquire brain signal control and the characteristics of their brain signal during the tasks that the stroke participants attempted.

ELIGIBILITY:
Inclusion Criteria:

* medically stable and >/= 6 months post stroke
* difficulty using upper limb for functional tasks
* >21 years old

Exclusion Criteria:

* chronic, progressive medical condition (i.e. Parkinson's disease)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
EEG (electroencephalography) | Week 12
  measures brain activity during a specified movement task

CONTACTS AND LOCATIONS:
Overall Officials: Janis J Daly, PhD, MS, Principal Investigator — Malcom Randall VA Medical Center
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States